CLINICAL TRIAL: NCT06893107
Title: Assessment of Treatment Outcomes and Alveolar Bone Changes Following Intentional Replantation of Hopeless Periodontally Involved Single-Rooted Teeth - A Pre-test, Post-test Interventional Study
Brief Title: Study on Treatment Results and Bone Changes After Replanting Severely Affected Teeth - A Before-and-After Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fujairah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USTFREC2024-03-3
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis; Periodontally compromised tooth; Intentional replantation
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: This study follows a single-group assignment model where all participants undergo intentional replantation of hopeless periodontally involved single-rooted teeth. It uses a pre-test, post-test design, with assessments at two time points. At baseline, CBCT and clinical exams assess alveolar bone levels, periapical status, and periodontal condition. The intervention involves careful extraction, conditioning, replantation, and stabilization of the tooth. A follow-up CBCT scan at 9 months evaluates changes in alveolar bone levels, root resorption, and periodontal healing. Clinical evaluations assess tooth stability, periodontal health, and patient-reported outcomes. Key outcomes include bone height, resorption, and periodontal healing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intentional Replantation of Hopeless Periodontally Involved Single-Rooted Teeth (Experimental): This study evaluates the outcomes of intentional replantation of hopeless periodontally involved single-rooted teeth using a pre-test, post-test interventional design.
  At baseline, clinical and CBCT assessments will be performed to evaluate alveolar bone levels, periodontal status, and tooth mobility. The intervention involves atraumatic extraction, extraoral conditioning (if needed), and replantation with stabilization.
  At 9 months, follow-up CBCT and clinical evaluations will assess bone changes, periodontal healing, and tooth stability.
  Interventions: Procedure: Intentional Replantation

INTERVENTIONS:
Procedure: Intentional Replantation — The intervention involves intentional replantation (IR) of periodontally compromised single-rooted teeth. Patients are selected based on criteria ensuring no vertical root fractures and potential for restoration. Preoperative preparation includes radiographic evaluation (CBCT/periapical), scaling, and root planing, along with antibiotic prophylaxis. The tooth is extracted non-traumatically using periotomes to preserve the periodontal ligament (PDL). After extraction, the tooth is stored in a sterile medium and granulation tissue is excised. Optional modifications (apical resection, retrograde filling, or surface treatment) may be performed. The tooth is then replanted into the socket, secured with a non-rigid splint, and occlusal adjustment is made. Postoperative care includes analgesics, antibiotics, and chlorhexidine rinse. Follow-ups are scheduled at 1 week, 4 weeks, and 9 months for evaluation of healing, survival, and patient-reported outcomes.

SUMMARY:
This research aims to evaluate the effectiveness of intentional replantation (IR) as a treatment for single-rooted teeth diagnosed as hopeless due to true periodontic lesions. The study will assess changes in alveolar bone and periodontal tissues, symptom resolution, and patient-reported outcomes (satisfaction and quality of life) following the procedure. Cone beam computed tomography (CBCT) imaging will be used to track radiographic changes at baseline and 9 months, while clinical examinations will monitor symptom resolution, including pain, swelling, and tooth mobility.

The study is a single-arm pre-test, post-test interventional design conducted at the College of Dentistry, University of Science and Technology Fujairah (new name: University of Fujairah). Participants will include adults aged 18-70 with single-rooted teeth deemed hopeless due to periodontic lesions. Participants will undergo intentional replantation, and data will be collected through clinical examinations, radiographic images, and patient questionnaires at baseline and 9 months.

Statistical analysis will compare pre- and post-treatment outcomes using paired-samples t-tests or Wilcoxon signed-rank tests, depending on data normality. The study aims to provide a comprehensive evaluation of intentional replantation, contributing valuable insights into its clinical effectiveness for managing complex dental conditions.

DETAILED DESCRIPTION:
The intervention in this study is intentional replantation (IR) of periodontally compromised single-rooted teeth deemed hopeless. Patients are chosen according to specific criteria, ensuring that the teeth are amenable to restoration and devoid of vertical root fractures. Preoperative preparation entails radiographic evaluation via periapical or cone-beam computed tomography (CBCT), scaling and root planing, and antibiotic prophylaxis when warranted. The process commences with a non-traumatic extraction utilising periotome to maintain the integrity of the periodontal ligament (PDL). After extraction, the tooth is handled extraorally within 15 minutes to preserve periodontal ligament viability. It is preserved in a sterile medium, such as saline or blood, and granulation tissue is meticulously excised. Optional root modifications, such as apical resection, retrograde filling with mineral trioxide aggregate or biodentine, or surface treatment with tetracycline or enamel matrix derivatives like Emdogain, may be conducted if required. The tooth is subsequently replanted into its original socket and secured with a non-rigid splint (fiber-reinforced composite or orthodontic wire) for a duration of 2 to 4 weeks. Occlusal adjustment is conducted to reduce excessive functional forces. Postoperative care comprises analgesics, antibiotics as necessary, and a 0.12% chlorhexidine rinse administered bi-daily for a duration of two weeks. Patients are instructed to adhere to a soft diet for two weeks to avert trauma to the replanted tooth. Follow-up evaluations are planned at 1 week, 4 weeks, 9 months to evaluate healing, bone regeneration, periodontal reattachment, and overall tooth viability. The principal outcome measures encompass tooth survival, periodontal healing, and bone regeneration, whereas secondary outcomes evaluate patient-reported pain, functionality, and quality of life.

In this study, the comparator is the tooth's pre-treatment condition, which serves as the baseline for comparison. Given that the study used a pre-test, post-test interventional design, each tooth serves as its own control. Baseline examinations, encompassing clinical indicators (mobility, probing depth, gingival inflammation) and radiographic evaluation (bone level, periodontal ligament space, root resorption), are documented prior to intentional replantation. Subsequent to the intervention, these measures are reassessed at 9-month follow-up to evaluate treatment outcomes and alterations in alveolar bone. This comparison facilitates an impartial assessment of the efficacy of purposeful replantation in enhancing periodontal health and bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the specified criteria will be included in the study.

* The patients with American Society of Anesthesiologists physical status classification 1 and 2.
* Radiographic bone loss of at least 50% around the targeted tooth.
* Probing depth of at least 5 millimetres around the targeted tooth.
* Grade III mobility (extreme mobility) of the targeted tooth according to Miller's classification.
* Grade II mobility or less (minimal to slight increased mobility without functional impairment) of adjacent teeth.
* Distance between the targeted tooth and adjacent teeth less than 2 millimetres.
* Patient preference for tooth retention through intentional replantation over extraction.

Exclusion Criteria:

* Previous history of failed IR.
* Severe anatomical limitations in the treatment area.
* Unwillingness to adhere to follow-up protocols

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Success of IR procedure | Baseline and 9 months post-replantation
  Definition: Success will be assessed based on clinical and radiographic outcomes at 9 months post-replantation.
  Key indicators:
  Preservation of alveolar bone levels (measured via CBCT and periapical radiographs).
  Absence of significant root resorption. Re-establishment of periodontal ligament attachment around the replanted tooth. Unit of Measurement: Binary outcome (Success vs. Failure)

SECONDARY OUTCOMES:
Change in Pain Level | Baseline and 9 months post-replantation
  Definition: Pain level will be assessed using the Visual Analog Scale (VAS), which ranges from 0 (no pain) to 10 (unbearable pain).
  Unit of Measurement: VAS score (0-10)
Change in Tooth Mobility | Baseline and 9 months post-replantation
  Definition: Tooth mobility will be measured using Miller's Mobility Criteria (Grade 0-3). Where 0 indicates No mobility. 3 indicates movement of more than 1 mm in horizontal direction with mobility in the vertical direction OR movement of more than 2 mm in Horizontal direction OR vertical mobility Unit of Measurement: Mobility grade (ordinal scale: 0-3)
Change in Probing Depth (PD) | Baseline and 9 months post-replantation
  Definition: Probing Depth will be measured using a WHO periodontal probe at four surfaces (mesial, distal, buccal, lingual).
  Unit of Measurement: Probing Depth (millimeters, mm)
Change in Bleeding on Probing (BOP) | Baseline and 9 months post-replantation
  Definition: Bleeding on Probing (BOP) will be recorded as present or absent. Unit of Measurement: Bleeding on Probing (Binary: Present/Absent)
Change in Alveolar Bone Loss Percentage (BL%) | Baseline and 9 months post-replantation
  Definition: BL% will be calculated using the formula:
  BL%= (L-Lr)/L ×100, where L = total root length, and Lr = remaining alveolar bone height.
  Unit of Measurement: Percentage (%)
Change in Oral Health-Related Quality of Life (OHRQoL) | Baseline and 9 months post-replantation
  Definition: Assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire.
  Unit of Measurement: OHIP-14 score (range: 0-56, higher scores indicate worse quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Nabeel Ayappali Kalluvalappil, MDS, Principal Investigator — Lecturer, College of Dentistry, University of Fujairah, UAE, Zip Code 2202
Locations (1):
- Dental Clinic, College of Dentistry, University of Fujairah,, Fujairah, Emirate of Fujairah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers. Data will only be used for analysis within the scope of this study and will not be publicly available.

REFERENCES:
- [Result] Praveen Kumar V, Sadasiva K, Raj Kumar J, Ramachandran A, Parthasarathy R, Thanikachalam Y. Current Trends in Intentional Replantation Treatment Among Endodontists and Postgraduate Students in India, the United States of America, and the United Kingdom: A Cross-Sectional Study. Cureus. 2023 May 30;15(5):e39742. doi: 10.7759/cureus.39742. eCollection 2023 May. PMID 37398781
- [Result] Pisano M, Di Spirito F, Martina S, Sangiovanni G, D'Ambrosio F, Iandolo A. Intentional Replantation of Single-Rooted and Multi-Rooted Teeth: A Systematic Review. Healthcare (Basel). 2022 Dec 21;11(1):11. doi: 10.3390/healthcare11010011. PMID 36611471
- [Result] Cunliffe J, Ayub K, Darcey J, Foster-Thomas E. Intentional replantation - a clinical review of cases undertaken at a major UK dental school. Br Dent J. 2020 Aug;229(4):230-238. doi: 10.1038/s41415-020-1988-6. PMID 32855480
- [Result] Becker BD. Intentional Replantation Techniques: A Critical Review. J Endod. 2018 Jan;44(1):14-21. doi: 10.1016/j.joen.2017.08.002. Epub 2017 Oct 21. PMID 29033086
- [Result] Mainkar A. A Systematic Review of the Survival of Teeth Intentionally Replanted with a Modern Technique and Cost-effectiveness Compared with Single-tooth Implants. J Endod. 2017 Dec;43(12):1963-1968. doi: 10.1016/j.joen.2017.08.019. Epub 2017 Oct 20. PMID 29061358
- [Result] Asgary S, Talebzadeh B. Intentional replantation of a molar with several endodontic complications. J Stomatol Oral Maxillofac Surg. 2019 Nov;120(5):489-492. doi: 10.1016/j.jormas.2018.11.019. Epub 2018 Dec 7. PMID 30529534
- [Result] Cho SY, Lee SJ, Kim E. Clinical Outcomes after Intentional Replantation of Periodontally Involved Teeth. J Endod. 2017 Apr;43(4):550-555. doi: 10.1016/j.joen.2016.11.024. Epub 2017 Feb 16. PMID 28215343
- [Result] Wang L, Jiang H, Bai Y, Luo Q, Wu H, Liu H. Clinical outcomes after intentional replantation of permanent teeth: A systematic review. Bosn J Basic Med Sci. 2020 Feb 5;20(1):13-20. doi: 10.17305/bjbms.2019.3937. PMID 30684952
- [Result] Zhang J, Luo N, Miao D, Ying X, Chen Y. Intentional replantation of periodontally involved hopeless teeth: a case series study. Clin Oral Investig. 2020 May;24(5):1769-1777. doi: 10.1007/s00784-019-03039-z. Epub 2019 Aug 13. PMID 31410671
- [Result] Park SH, Paek SH, Kim B, Lee JT. Assessment of Bone Height Changes Based on the Cone-Beam Computed Tomography Following Intentional Replantation for Periodontally Compromised Teeth. Medicina (Kaunas). 2022 Dec 25;59(1):40. doi: 10.3390/medicina59010040. PMID 36676664
- [Derived] Ayappali Kalluvalappil N, Kumar RS, Hassan TH. Intentional replantation of periodontally compromised teeth with concentrated growth factors. Clin Adv Periodontics. 2025 Oct 14. doi: 10.1002/cap.70017. Online ahead of print. PMID 41085111